CLINICAL TRIAL: NCT05382910
Title: Phase Ib/II Clinical Trial of Safety, Pharmacokinetics and Preliminary Efficacy of MG-K10 Humanized Monoclonal Antibody Injection in Adult Asthmatic Subjects
Brief Title: A Study of MG-K10 in Subjects With Asthma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-K10-AS-2
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: About 180 subjects with moderate-to-severe asthma who meet the inclusion criteria will be selected for this study, according to 1:1:1 Randomly assigned to one of the MG-K10 Q2W group, the MG-K10 Q4W group, and the placebo group, with approximately 60 subjects in each group. The Q2W group will receive MG-K10 300mg subcutaneous injection every 2 weeks; Q4W group will receive MG-K10 300mg subcutaneous injection (every 4 weeks) + 2ml placebo subcutaneous injection ; the placebo group will receive 2 ml of placebo subcutaneously administered every 2 weeks. All three groups were followed up for 8 weeks after 24 weeks of treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MG-K10 Q2W (Experimental): Received MG-K10 300 mg subcutaneous injection every 2 weeks
  Interventions: Drug: MG-K10
- MG-K10 Q4W (Experimental): Received MG-K10 300 mg subcutaneous injection every 4 weeks
  Interventions: Drug: MG-K10; Drug: Placebo
- Placebo (Placebo Comparator): The placebo group will receive 2 ml of placebo subcutaneously administered every 2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MG-K10 — MG-K10 Humanized Monoclonal Antibody Injection
  Arms: MG-K10 Q2W; MG-K10 Q4W
Drug: Placebo — Placebo
  Arms: MG-K10 Q4W; Placebo

SUMMARY:
This study is a phase Ib/II clinical trial conducted in Chinese adult asthmatic subjects to evaluate the preliminary efficacy and safety of MG-K10 humanized monoclonal antibody injection in the treatment of asthma.

DETAILED DESCRIPTION:
The study was conducted in two phases: the Phase Ib study focused on the safety and tolerability of MG-K10 in adult asthma subjects. Phase II study focused on the preliminary efficacy in adults with moderate to severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed according to the 2021 version of the GINA guidelines for at least 1 year;
* 1 second forced expiratory volume (FEV1) before randomization before bronchodilator use The measured value is ≤80% of the normal predicted value;
* Must have experienced at least one severe acute asthma attack within 12 months outbreak event.
* Positive bronchodilator test
* Subjects and partners agree to take effective contraceptive measures from signing the Informed Consent Form (ICF) to 6 months after the end of treatment

Exclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease (COPD) or other lung diseases that may impair lung function
* Subjects with malignant tumor within 5 years
* Received biologics with the same therapeutic purpose within 6 months prior to screening,
* Women who are breastfeeding or pregnant, or who plan to become pregnant or breastfeeding during the study period;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Absolute Change from baseline in pre-bronchodilator FEV1 | 12 week
  Absolute change from baseline in pre-bronchodilator FEV1 in each study group at 12 week of MG-K10 treatment compared with placebo

SECONDARY OUTCOMES:
Absolute Change from baseline in pre-bronchodilator FEV1 | 4,8,16,20,24,28,32 week
  Absolute change from baseline in pre-bronchodilator FEV1 in each study group at 4,8,16,20,24,28,32 week of MG-K10 treatment compared with placebo
Percent change from baseline in pre-bronchodilator FEV1 | 4,8,16,20,24,28,32 week
  at 4,8,16,20,24,28,32 week of MG-K10 treatment compared with placebo，Percent change from baseline in pre-bronchodilator FEV1
peak morning and evening expiratory flow (PEF) | 4,8,12,16,20,24,28,32 week
  Change from peak morning and evening expiratory flow (PEF) compared with baseline (absolute and percentage)
the Annualized rate of severe asthma acute event | 24 weeks and 25 to 32 weeks
  The annualized rate of severe asthma acute event within 24 weeks and 25 to 32 weeks of treatment
Annualized rate of the event of loss of asthma control (LOAC) | 24 weeks and 25 to 32 weeks
  the annualized rate of the event of loss of asthma control (LOAC) at 24 weeks and 25 to 32 weeks of treatment
Time of the first severe asthma acute event | 32 weeks
  Time of the first severe asthma acute event
Time of first loss of asthma control (LOAC) | 32weeks
  Time of first loss of asthma control (LOAC)
asthma Control Questionnaire 5 (ACQ-5 score 0-30) changes in score | 4, 8, 12, 16, 20, 24, 28, and 32 weeks
  There are 5 questions in ACQ5, It is a questionnaire used to evaluate the degree of asthma control. Each question is scored from 0 to 6 (on a 7-point scale) according to its severity. The higher the score, the less satisfactory symptom control
Morning/evening asthma symptom score | 24 and 32 week
  Patients will record total symptom scores in morning（a 0-4 scale, with 0=no symptoms, 4=inability to fall asleep at night due to symptoms) and evening (a 0-4 scale, with 0=no symptoms, 4=severe symptoms, unable to work or perform daily activities)
Daily use of first aid medicine spray | 24 and 32 week
  Daily use of first aid medicine spray compared with baseline
Incidence of Adverse events (AEs) | 32 weeks
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing
Pharmacokinetic concentration | 32 weeks
  To evaluate the Pharmacokinetic concentration of MG-K10 for each dose group. Population pharmacokinetic analysis is performed using a nonlinear mixed-effects model
Fractional exhaled nitric oxide (FeNO) | 32 weeks
  At each evaluation time point, the changes of Fractional exhaled nitric oxide(FeNO) were compared with baseline in each group
thymus activation regulated chemokine (TARC) | 32 weeks
  At each evaluation time point, the changes of thymus activation regulated chemokine (TARC) were compared with baseline in each group
serum immunoglobulin E (IgE) | 32 weeks
  At each evaluation time point, the changes of serum immunoglobulin E (IgE)were compared with baseline in each group
Anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) | 32 weeks
  Incidence of anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, Medical PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No